CLINICAL TRIAL: NCT00454779
Title: A Randomized, Open-Label, Controlled, Phase II Trial of Combination Chemotherapy With or Without Panitumumab as First-line Treatment of Subjects With Metastatic or Recurrent Head and Neck Cancer, and Cross-over Second-line Panitumumab Monotherapy of Subjects Who Fail the Combination Chemotherapy…
Brief Title: PARTNER: Panitumumab Added to Regimen for Treatment of Head aNd Neck Cancer Evaluation of Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050236
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Metastatic or Recurrent Squamous Cell Carcinoma of Head and Neck
Keywords: SCCHNC; Metastatic; Recurrent
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence | interventions — Cisplatin; Panitumumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Panitumumab + Docetaxel + Cisplatin
  Interventions: Drug: Panitumumab; Drug: Cisplatin; Drug: Docetaxel
- Arm 2 (Other): control
  Interventions: Drug: Cisplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Cisplatin — chemotherapy arm
  Arms: Arm 2
Drug: Panitumumab — experimental arm
  Arms: Arm 1
Drug: Docetaxel — chemotherapy arm
  Arms: Arm 2
Drug: Cisplatin — experimental arm
  Arms: Arm 1
Drug: Docetaxel — experimental arm
  Arms: Arm 1

SUMMARY:
This is a randomized, open-label, 2-arm, controlled, phase 2, multi-center, estimation clinical trial of docetaxel and cisplatin combination chemotherapy with and without panitumumab in the first-line treatment of subjects with metastatic or recurrent head and neck cancer, as well as a cross-over second-line panitumumab monotherapy of subjects who fail the chemotherapy only arm. This study will be conducted in the United States. Approximately 150 subjects with histologically or cytologically confirmed metastatic and/or recurrent SCCHN.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic and/or recurrent Squamous Cell Carcinoma of Head and Neck (SCCHN) determined to be incurable by surgery and/or radiation therapy.
* Measurable disease by CT scan
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
* Age: 18 years or older
* Adequate hematologic, renal, metabolic, hepatic & thyroid function

Exclusion Criteria:

* Prior systemic treatment for metastatic and/or recurrent SCCHN
* CNS metastases, or nasopharyngeal carcinoma
* History of interstitial lung disease
* History of another primary cancer
* Any co-morbid disease that would increase risk of toxicity

  * Active infection requiring systemic treatment
  * Prior anti-Epidermal Growth Factor receptor (anti-EGFr) antibody therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2012-06-11 (Actual); Study Completion 2014-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (102):
- United States (70):
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, La Verne, California
  - Research Site, Los Angeles, California
  - Research Site, Santa Cruz, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Norwich, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Orlando, Florida
  - Research Site, Athens, Georgia
  - Research Site, Griffin, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Centralia, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Zion, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Ashland, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Pascagoula, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Jefferson City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Hackensack, New Jersey
  - Research Site, Binghamton, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Nyack, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Scranton, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Galveston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Chesapeake, Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Marshfield, Wisconsin
- Austria (4):
  - Research Site, Graz
  - Research Site, Leoben
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (7):
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Kortrijk
  - Research Site, Libramont
  - Research Site, Liège
  - Research Site, Ottignies
  - Research Site, Wilrijk
- Czechia (3):
  - Research Site, Brno
  - Research Site, Prague
  - Research Site, Znojmo
- France (4):
  - Research Site, Angers
  - Research Site, Lens
  - Research Site, Perpignan
  - Research Site, Vandœuvre-lès-Nancy
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Research Site, San Juan, Puerto Rico
- Slovakia (5):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Nové Zámky
  - Research Site, Prešov
  - Research Site, Spišská Nová Ves
- Spain (6):
  - Research Site, Santander, Cantabria
  - Research Site, Barcelona, Catalonia
  - Research Site, Girona, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid

REFERENCES:
- [Background] Wirth LJ. PARTNER: a study of panitumumab plus chemotherapy for first-line treatment of advanced head and neck cancer. Commun Oncol. 2008;5(Supp 14):1-4.
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 29 January 2007 to 1 September 2010.
Pre-assignment Details: The planned number of subjects to enroll was 110. The actual number of subjects enrolled was 113.
Groups:
- Panitumumab Plus Chemotherapy: Panitumumab + Docetaxel + Cisplatin, experiment
- Chemotherapy Alone: Docetaxel + Cisplatin, control
Period: First-line Treatment Phase
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Started | 56 | 57
Received Study Medication | 56 | 55
Completed | 51 (Disease progression (radiographically determined) or death) | 49 (Disease progression (radiographically determined) or death)
Not Completed | 5 | 8
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Ended follow-up prior to analysis | 1 | 1
Not completed — Ongoing | 1 | 0
Period: Second-line Treatment Phase
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Started | 0 (Subjects in this arm do not have second-line treatment period) | 30 (Second-line Panitumumab Monotherapy)
Completed | 0 (Disease progression (radiographically determined) or death) | 27 (Disease progression (radiographically determined) or death)
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Ended follow-up prior to analysis | 0 | 1
Not completed — Ongoing | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (8.6) | 58.9 (7.4) | 58.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 47 | 52 | 99

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) During the First-line Treatment Phase
Description: The time from the date of randomization to the date of first disease progression determined by the investigators per modified RECIST v1.0, or death within 60 days after the last evaluable tumor assessment or randomization date (whichever is later) during the first-line treatment phase.
Time Frame: Every 6 weeks until disease progression or death, up to 67 months
Population: All randomized participants < 70 years of age who provide informed consent and receive at least one dose of first-line treatment (chemotherapy and/or panitumumab)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 52 | 51
Months | 6.9 [4.7 to 8.3] | 5.5 [4.1 to 6.8]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; p = 0.051, Regression, Cox; Stratified by IVRS randomization factors; Hazard Ratio (HR) = 0.629, 95% CI 2-sided [0.395 to 1.002] — Hazard ratio is presented as panitumumab plus chemotherapy:chemotherapy alone
Statistical Analysis 2: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; p = 0.048, Log Rank; Stratified by IVRS randomization factors

2. Secondary Outcome: Overall Response Rate (ORR) During the First-line Treatment Phase
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (SLD) of target lesions from baseline; Overall Response (OR) = CR + PR. An overall response of CR or PR must be confirmed at least 4 weeks after the criteria for response are first met. ORR is the percentage of subjects with an overall response among the analysis population.
Time Frame: Every 6 weeks until disease progression or death, up to 67 months
Population: all randomized subjects < 70 years of age who provide informed consent and receive at least one dose of first-line treatment (chemotherapy and/or panitumumab), with at least one uni-dimensionally measurable lesion at baseline using a modified RECIST v1.0 per investigators' review
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 52 | 51
Percentage of Participants | 44.23 [30.73 to 57.73] | 37.25 [23.99 to 50.52]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; Mean Difference (Final Values) = 6.23, 95% CI 2-sided [-11.67 to 24.12] — With Mantel-Haenszel weights within strata defined by randomization factors recorded in the IVRS
Statistical Analysis 2: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; Odds Ratio (OR) = 1.37, 95% CI [0.57 to 3.33] — Calculated from a logistic regression model with treatment indicator and randomization factors (recorded on the CRF) as covariates

3. Secondary Outcome: Rate of Disease Control (RDC) During the First-line Treatment Phase
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (SLD) of target lesions from baseline; Disease Progression (PD), >=20% increase in the SLD of target lesions from nadir; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. An overall response of CR or PR must be confirmed at least 4 weeks after the criteria for response are first met. A best overall response of SD requires a visit response of SD or better no earlier than 35 days after randomization. RCD is the percentage of subjects with a best overall response of CR, PR or SD among the analysis population.
Time Frame: Every 6 weeks until disease progression or death, up to 67 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 52 | 51
Percentage of Participants | 80.77 [70.06 to 91.48] | 72.55 [60.30 to 84.80]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; Mean Difference (Final Values) = 7.78, 95% CI 2-sided [-8.29 to 23.85] — With Mantel-Haenszel weights within strata defined by randomization factors recorded in the IVRS
Statistical Analysis 2: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; Odds Ratio (OR) = 1.76, 95% CI [0.62 to 5.26] — [estimate comment as in outcome 2, analysis 2]

4. Secondary Outcome: Duration of Response (DOR) During the First-line Treatment Phase
Description: Calculated only for the subset of subjects who have an overall response of CR or PR while on first-line treatment phase (subsequently confirmed at least 4 weeks thereafter), and is defined as time from the first CR or PR to the first observed disease progression by a modified RECIST v1.0. Subjects not meeting the criteria for progression by the analysis data cutoff date will be censored at their last evaluable disease assessment date.
Time Frame: Every 6 weeks until disease progression or death, up to 67 months
Population: All randomized participants < 70 years of age who provide informed consent and receive at least one dose of first-line treatment (chemotherapy and/or panitumumab), with at least one uni-dimensionally measurable lesion at baseline using a modified RECIST v1.0 per investigators' review and objective response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 23 | 19
Months | 8.0 [5.7 to 11.1] | 5.1 [4.4 to 7.2]

5. Secondary Outcome: Time to Response (TTR) During the First-line Treatment Phase
Description: Time from the date of randomization to the first CR or PR during first line treatment phase (subsequently confirmed at least 4 weeks thereafter)
Time Frame: Every 6 weeks until disease progression or death, up to 67 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 23 | 19
Weeks | 8.8 (3.9) | 10.6 (6.1)

6. Secondary Outcome: Overall Survival (OS) for the First-line Treatment
Description: Time from the date of randomization to the date of death during the entire study
Time Frame: Until death, up to 67 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 52 | 51
Months | 12.9 [9.4 to 18.5] | 13.8 [11.8 to 22.9]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; p = 0.663, Regression, Cox; Stratified by IVRS randomization factors; Hazard Ratio (HR) = 1.103, 95% CI 2-sided [0.709 to 1.717] — Hazard ratio is presented as panitumumab plus chemotherapy:chemotherapy alone
Statistical Analysis 2: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; p = 0.666, Log Rank; Stratified by IVRS randomization factors

7. Secondary Outcome: Progression Free Survival (PFS) During the Second-line Treatment Phase
Description: The time from the first dose of panitumumab monotherapy to the date of first disease progression determined by the investigators per modified RECIST v1.0, or death within 60 days after the last evaluable tumor assessment or the second-line first dose date (whichever is later) during the second-line treatment phase.
Time Frame: Every 6 weeks until disease progression or death, up to 57 months
Population: Subjects who are randomized to docetaxel and cisplatin chemotherapy alone treatment for their first-line treatment and treated subsequently with at least 1 dose of second-line panitumumab monotherapy
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 0 | 30
Months |  | 4.2 [1.5 to 7.6]

8. Secondary Outcome: Overall Response Rate (ORR) During the Second-line Treatment Phase
Description: as for outcome 2
Time Frame: Every 6 weeks until disease progression or death, up to 57 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 0 | 30
Percentage of Participants |  | 13.33 [1.17 to 25.50]

9. Secondary Outcome: Rate of Disease Control (RDC) During the Second-line Treatment Phase
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (SLD) of target lesions from baseline; Disease Progression (PD), >=20% increase in the SLD of target lesions from nadir; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. An overall response of CR or PR must be confirmed at least 4 weeks after the criteria for response are first met. A best overall response of SD requires a visit response of SD or better no earlier than 35 days after the first dose date in second-line treatment. RCD is the percentage of subjects with a best overall response of CR, PR or SD among the analysis population.
Time Frame: Every 6 weeks until disease progression or death, up to 57 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 0 | 30
Percentage of Participants |  | 53.33 [35.48 to 71.19]

10. Secondary Outcome: Duration of Response (DOR) During the Second-line Treatment Phase
Description: Time from the first CR or PR to the first observed disease progression by a modified RECIST v1.0. Subjects not meeting the criteria for progression by the analysis data cutoff date will be censored at their last evaluable disease assessment date.
Time Frame: Every 6 weeks until disease progression or death, up to 57 months
Population: Subjects who are randomized to docetaxel and cisplatin chemotherapy alone treatment for their first-line treatment and treated subsequently with at least 1 dose of second-line panitumumab monotherapy, with at least one uni-dimensionally measurable lesion at baseline using a modified RECIST v1.0 per investigators' review and objective response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 0 | 4
Months |  | NA [5.1 to NA] — Median is not reached due to censoring.

11. Secondary Outcome: Time to Response (TTR) During the Second-line Treatment Phase
Description: Time from the first dose of panitumumab monotherapy to the first CR or PR during second-line treatment phase (subsequently confirmed at least 4 weeks thereafter)
Time Frame: Every 6 weeks until disease progression or death, up to 57 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 0 | 4
Weeks |  | 10.6 (5.6)

12. Secondary Outcome: Overall Survival (OS) for the Second-line Treatment
Description: Time from the first dose of panitumumab monotherapy to the date of death during the entire study
Time Frame: Until death, up to 57 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 0 | 30
Months |  | 8.5 [6.5 to 13.2]

ADVERSE EVENTS:
Time Frame: The time frame for adverse event reporting is from the first dose date to 30 days since the last dose date of the first-line treatment. The median time frame is 4.5 months for Panitumumab Plus Chemotherapy arm and 4.4 months for Chemotherapy Alone arm.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Serious Adverse Events (participants affected / at risk) | 34/56 | 27/55
Other Adverse Events (participants affected / at risk) | 54/56 | 53/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Chemotherapy (N=56) | Chemotherapy Alone (N=55)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Aphagia (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4
Oral cavity fistula (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Device dislocation (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 3 | 0
Localised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 4
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 6
Pneumonia staphylococcal (Infections and infestations) | 2 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 3
Renal failure acute (Renal and urinary disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Chemotherapy (N=56) | Chemotherapy Alone (N=55)
Anaemia (Blood and lymphatic system disorders) | 22 | 27
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 7 | 5
Neutropenia (Blood and lymphatic system disorders) | 9 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5
Tinnitus (Ear and labyrinth disorders) | 0 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 4
Conjunctivitis (Eye disorders) | 8 | 0
Lacrimation increased (Eye disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 15 | 9
Diarrhoea (Gastrointestinal disorders) | 25 | 16
Dry mouth (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 6
Dysphagia (Gastrointestinal disorders) | 9 | 4
Mouth ulceration (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 34 | 33
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 9 | 3
Vomiting (Gastrointestinal disorders) | 15 | 18
Asthenia (General disorders) | 13 | 5
Chills (General disorders) | 5 | 3
Face oedema (General disorders) | 4 | 1
Fatigue (General disorders) | 28 | 28
Mucosal inflammation (General disorders) | 15 | 7
Oedema (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 4 | 10
Pain (General disorders) | 4 | 1
Pyrexia (General disorders) | 8 | 8
Bronchitis (Infections and infestations) | 3 | 1
Candidiasis (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 0
Haemoglobin decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 13 | 11
Cachexia (Metabolism and nutrition disorders) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 20 | 10
Dehydration (Metabolism and nutrition disorders) | 11 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 23 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 13 | 7
Dysgeusia (Nervous system disorders) | 5 | 6
Headache (Nervous system disorders) | 5 | 8
Neuropathy peripheral (Nervous system disorders) | 9 | 11
Paraesthesia (Nervous system disorders) | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 5
Somnolence (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 8 | 6
Depression (Psychiatric disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 5 | 4
Nocturia (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acne (Skin and subcutaneous tissue disorders) | 7 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 14
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 13 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 3
Erythema (Skin and subcutaneous tissue disorders) | 7 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 21 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.